CLINICAL TRIAL: NCT02072109
Title: Evaluation of Regional Splanchnic Tissue Oxygenation Measured by NIRS (Near Infrared Spectroscopy) in Preterm Infants Receiving Bolus Versus Continuous Feeding
Brief Title: Comparison of Regional Splanchnic Tissue Oxygenation Measured by NIRS in Preterm Babies Fed Bolus Versus Continuous Feeding
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 267-13
Record Dates: First submitted 2014-02-24; First posted 2014-02-26 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2014-06

CONDITIONS: Premature; Infant, Light-for-dates; Feeding Patterns
Keywords: Near infrared spectroscopy; Bolus nutrition; Continuous nutrition; Mesenteric circulation
MeSH Terms: conditions — Premature Birth; Feeding Behavior

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Bolus feeding: Preterm infants born in Meir Medical Center and being treated in the Neonatal Intensive Care Unit
- Continuous feeding: Preterm infants born in Meir Medical Center and being treated in the Neonatal Intensive Care Unit

SUMMARY:
Early initiation of enteral feeding, achievement of full enteral feeding and cessation of parenteral nutrition are extremely important in the very premature infant. This way it is possible to achieve good post-natal growth and developement while minimizing the metabolic and infectious complications of parenteral feeding.

There isn't much information in literature regarding the impact of enteral feeding on intestinal blood flow and intestinal regional oxygenation in the preterm infant. There is also no consensus regarding the best regimen of delivering the enteral nutrition - bolus feeding or continuous feeding.

The aim of our study is to compare the intestinal regional oxygenation before and after two feeding regimens - bolus feeding and continuous feeding - in clinically stable preterm infants born before 32 weeks gestation. The evaluations will be performed using NIRS technology (Near Infrared Spectroscopy).

The study may help to assess which feeding regimen is gentler to the immature intestines (i.e. alters less the splanchnic blood flow and oxygenation) and therefore the preferred way to feed preterm infants.

DETAILED DESCRIPTION:
Early initiation of enteral feeding, achievement of full enteral feeding and cessation of parenteral nutrition are extremely important in the very premature infant. This way it is possible to achieve good post-natal growth and developement while minimizing the metabolic and infectious complications of parenteral feeding.

There isn't much information in literature regarding the impact of enteral feeding on intestinal blood flow and intestinal regional oxygenation in the preterm infant. There is also no consensus regarding the best regimen of delivering the enteral nutrition - bolus feeding or continuous feeding.

The aim of our study is to compare the intestinal regional oxygenation before and after two feeding regimens - bolus feeding and continuous feeding - in clinically stable preterm infants born before 32 weeks gestation. The evaluations will be performed using NIRS technology (Near Infrared Spectroscopy).

The investigators intend to assess 20 clinically stable, appropriate for gestational age preterm infants, born before 32 weeks of gestation and receiving full enteral feedings at least 1 week prior to enrollment with no signs of feeding intolerance.

All 20 participants evaluated constitute the 2 study groups:

1. Group 1 = Bolus feeding - before and after one bolus feeding
2. Group 2 = Continuous feeding - before and after one continuous feeding.

The study may help to assess which feeding regimen is gentler to the immature intestines (i.e. alters less the splanchnic blood flow and oxygenation) and therefore the preferred way to feed preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* Born 23+0 to 31+6 weeks gestational age.
* Appropriate for gestational age.
* Clinically stable.
* Full enteral feeding at least 1 week prior to enrollment.
* Bolus feeding.
* No signs of feeding intolerance.

Exclusion Criteria:

* Major congenital anomalies (severe heart or cerebral disease, chromosomal abnormalities, any malformation or disease of the gastrointestinal tract).
* Previous diagnosis of necrotizing enterocolitis or spontaneous intestinal perforation.
* Need for blood transfusion 1 week prior to enrollment.
* Need for vasopressor therapy 1 week prior to enrollment.
* Cutaneous disease not allowing the placement of the NIRS probe.

Ages: 10 Days to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm infants born in Meir Medical Center and being treated in the Neonatal Intensive Care Unit.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-02 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Change in splanchnic regional tissue oxygenation before and after a bolus / continuous feeding. | 10 hours
  Measurement of the regional tissue oxygenation of the intestines using NIRS (Near Infra-Red Spectroscopy) technology before and after a bolus feeding and then a continuous feeding.

CONTACTS AND LOCATIONS:
Overall Officials: Gisela Sirota, M.D., Principal Investigator — Meir Medical Center
Locations (1):
- Neonatal Intensive Care Unit - Meir Medical Center, Kfar Saba, Israel